CLINICAL TRIAL: NCT05214313
Title: Impact of a Standardized Music Therapy Protocol on the Quality of Life of Patients With Abnormal Movements Treated With Continuous Electrical Neuromodulation (Music-QOL)
Brief Title: Impact of a Standardized Music Therapy Protocol on the Quality of Life of Patients With Abnormal Movements Treated With Continuous Electrical Neuromodulation
Acronym: Music-QOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: investigator decision
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RECHMPL20_0672
Record Dates: First submitted 2022-01-05; First posted 2022-01-28 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Dystonia; Parkinson Disease; Essential Tremor
Keywords: Music therapy; Abnormal movements; Quality of life; Functional neurosurgery
MeSH Terms: conditions — Dystonia; Parkinson Disease; Essential Tremor; Dyskinesias | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Music therapy Intervention" group (G1) (Experimental): Patients in the "Music therapy intervention" group will also perform the 1st session of the program during the inclusion visit (V0). The patients will benefit from fourteen 1-hour music therapy sessions (15 min of reception, installation and debriefing at the end of the session and 45 min of program). The 14 individual sessions will be spread over three months at the rate of 2 weekly sessions the first month then a single weekly session the following month and finally 2 monthly sessions the last month. Patients will be assessed at inclusion, then the first month (V1) and at the end of the intervention (V2).
  Interventions: Behavioral: Music Therapy
- " Control " group (G2) (No Intervention): The patients in this group will benefit from the usual care corresponding to a quarterly medical examination. The patients will be assessed on the day of inclusion (V0) and then during the routine three-month medical examination (V2). At the end of the study, these patients will be able to benefit from the same music therapy program, offered under the same operating conditions.

INTERVENTIONS:
Behavioral: Music Therapy — The standardised music therapy protocol of 45 minutes will include at each session :
  * 10 min of musical listening in a soothing environment (relaxation chair and reduced and coloured lighting) in sensory isolation (with headphones) and aimed at relaxation as a preamble to the active phase of the protocol
  * Active phase: (25 min)
  * 5 min of receptive music therapy linked to a given emotion, different at each session (joy, sadness, anger and fear) aimed at emotional management (feeling and distancing),
  * 20 minutes of active music therapy with instrumental and vocal improvisation that solicits the body physiologically,
  * 10 minutes of musical listening in sensory isolation for a state of rest.
  The entire protocol is carried out with the permanent perception of heartbeats set to a physiological frequency of 50 to 100 BPM.
  Arms: "Music therapy Intervention" group (G1)

SUMMARY:
The study of the impact of music on emotional, motor and cognitive aspects remains recent. Music therapy has experienced a major boom over the last half century thanks to neuroradiological techniques for investigating the brain, and in particular in vivo functional MRI. Brain imaging has also made it possible to highlight and analyse certain activations of the networks concerned during the passive listening of music (receptive music therapy) but also during the playing of a musical instrument and/or the use of the voice (active music therapy). The accumulated data in music neurophysiology is now considerable [1]. Music therapy has thus been associated with motor rehabilitation in the case of acquired (stroke) and/or degenerative (Parkinson's disease) pathologies and has also been proposed as a means of pain relief. However, although proposed in the middle of the 20th century as a potentially therapeutic tool, music therapy has not managed to prove sufficiently effective to be validated in medicine. One of the limitations remains the intervention of numerous subjective factors, notably in the establishment of "protocols" and the absence of standardisation in their very structures.

Each year, the "Resistant Brain Pathology" unit of the Department of Neurosurgery takes care of more than a hundred patients who have benefited from treatment with Continuous Electrical Neuromodulation (CEN) in order to respond to a motor symptomatology that is resistant to the usual treatments. The benefits of DBS in the management of abnormal movements have been demonstrated [2]. However, this symptomatic treatment does not exclude a worsening of the underlying pathology over time, thereby increasing latent anxiety and promoting the fragility of otherwise severely disabled patients. The management of chronic diseases requires the expertise of a multidisciplinary team so that each aspect contributing to the quality of life of patients can be assessed and supported as best as possible.

In order to improve the quality of life of our patients, a music therapy unit has been established within the multidisciplinary neurosurgery department for two years now. The clinical music therapist attached to the unit has a dedicated room, offering a sensory environment conducive to relaxation and including all the necessary comfort. A standardised protocol for the conduct of the sessions, the organisation and choice of music in direct relation to the different emotions explored on the basis of the permanent perception of heartbeats was developed on the basis of the Webb & all study [3]. When a patient is immersed in a sound bath, identical to that perceived in utero, it would seem that this potentiates the benefits expected from music therapy sessions [3].

Our approach, although empirical, shows a decrease in anxiety and an increase in well-being in about fifty patients. Our observations support those highlighted in the literature in other pathologies [4] and encourage the use of this approach as a preamble to more specific explorations, in particular the catalysis of certain motor behaviours.

This project is therefore in line with this approach and continuity.

The investigators thus hypothesize that participation in a standardized music therapy protocol (active, receptive and psychomusical relaxation) against a background of regular heartbeats improves the quality of life of the operated patients by acting in particular on a reduction of anxiety and depressive symptoms.

To our knowledge, music therapy has never been proposed in a standardised way to patients with multiple disabilities, operated on and cared for over the long term in a functional neurosurgery department. This approach remains non-invasive and attractive in an often anxiety-provoking hospital context.

DETAILED DESCRIPTION:
Methodology:

This is a prospective, controlled, randomised, open-label, single-centre, two-arm, parallel, 1:1 ratio, non-drug therapeutic interventional study with three months of follow-up (Category 2)

The analysis of the primary and secondary endpoints will be conducted on an intention-to-treat (ITT) basis: each patient will be analysed in his or her randomisation arm once the patient has been assessed at inclusion and has received at least one assessment of the primary endpoint.

Initial comparability of groups A description of each group will be made by giving the frequencies of the different categories for the qualitative variables. As the distributions of the quantitative variables are not always Gaussian, the description of these variables will be done using the mean and the standard deviation but also the median and the minimum and maximum values. In case of non-comparability of the groups on one of the confounding factors, an adjustment or a stratification (in case of interaction) will be considered.

Analysis of primary endpoint The absolute change in the SF36 total score between the 2 assessments (T0 and T3 months) will be compared between the two groups using a Student's t test if the distribution is Gaussian or by a non-parametric test otherwise (Mann-Witney).

To estimate the "effect size", the variation of the score will be analysed by an analysis of covariance model including the intervention effect (ETP) and the SF36 inclusion value. In case of a non-Gaussian distribution, a transformation for normalisation will be applied and the normality of the residuals will be tested.

Analysis of secondary endpoints Changes in the SF36 score, SF36 subscores, anxiety and depression symptom scores and EVIBE will be analysed using the same methods as the primary endpoint.

Changes in knowledge of the disease will be analysed for each domain (Chi-2 test or Fisher's exact test) in intergroup and intragroup (Mac-Nemar's chi2) at 1 and 3 months.

Depending on the nominal, ordinal or continuous nature of the other clinical and socio-demographic variables, the analysis is carried out using Pearson's, Spearman's or Kendall's correlation coefficients, using a Chi-square test or Fisher's exact test, or using parametric (Student's or ANOVA) or non-parametric (Mann Whitney's and Kruskall Wallis' test) tests of comparison of means.

The alpha risk will be set at 5% for all tests. The statistical analysis will be carried out at the clinical research unit of the Department of Medical Information of the Montpellier CHRU with SAS version 9 software (SAS Institute, Cary, N.C.).

Number of patients:

The calculation of the number of subjects was carried out in collaboration with the Clinical and Epidemiological Research Unit of the University Hospital of Montpellier.

Based on the study [5] available in this field and using the SF36, the investigators hypothesise that the difference in variation of the total quality of life score (primary endpoint) to be highlighted between the 2 groups would be of the order of 10 points, with a standard deviation of 13. With a power of 80% and a first order risk of 5%, 27 subjects per group would be required. Anticipating a 10% drop-out rate, the number of patients to be recruited is 30 subjects in each arm, or 60 subjects in total.

Patient selection:

The patients likely to be included in the study are adults, followed in the functional neurosurgery department, associated with the "resistant brain pathology" unit, operated, treated by Continuous Electrical Neuromodulation, and medically stabilized.

Duration of project:

Duration of the inclusion period: 24 months Duration of participation of each participant: 3 months Duration of statistical analysis and final report writing: 7 months Expected duration of the study: 34 months

Schedule visit:

During a follow-up hospitalisation in the unit, patients will be systematically informed about the music therapy protocol. If the patients meet the inclusion criteria and agree to participate in our research, after signing the consent form with the study doctor, the patients will be called for an inclusion visit (V0). During this V0 visit, the patients will be received by the music therapist in order to carry out a psychomusical assessment of about 1 hour, then by the neuropsychologist to submit them to the various evaluations mentioned below.

Patients will then be randomised to one of two groups : "intervention" group or "control" group.

The music therapy programme will consist of 14 sessions spread over three months, with two weekly sessions in the first month, a single weekly session in the following month and two monthly sessions in the last month. Given the pilot nature of our study, the investigators will carry out an evaluation at 1 month (V1) in order to observe the impact of the protocol proposed intensively in the first month. A final evaluation will be proposed by the neuropsychologist at the end of the study. This will be coupled with a routine medical visit in the unit (V2).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years)
* Meets eligibility criteria: treated with CEN and medically stabilised

Exclusion Criteria:

* Not be available for 3 consecutive months
* Not be able to speak and understand the French language
* Severe disability that would prohibit musical practice according to the investigator (such as tetraparesis, anarthria...)
* Lack of informed consent
* Foreseeable absence from at least 30% of the sessions
* Pregnancy in progress or planned during the study, pregnant or breastfeeding
* Adult protected by law or patient under guardianship or curatorship
* Not residing in Occitania
* Not covered by a social security scheme
* Participation in another ongoing research project
* Complementary therapeutic treatment such as 3rd wave Cognitive Behavioural Therapy (mindfulness or relaxation type)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Change of total score of Quality of life assessment (MOS SF-36) baseline at 1 month and 3 months | The evaluations will take place at three times : at patient inclusion (V0), at 1 month (V1) and at 3 months from the intervention (V2).
  It is a generic scale, it can be administered to subjects with a wide range of health problems, or even to healthy subjects in the general population.The scale can be administered as a self-administered questionnaire or as a hetero-questionnaire and requires only 5 to 10 minutes.
  There are 11 questions in the SF-36, with 36 items in total. Its assess 8 dimensions divided into two: a physical component and a mental component.
  The ninth dimension consists of a single question: Evolution of perceived health.
  The patient assesses his or her current health status by comparing it to his or her health status one year earlier. This item provides an indicator of the change in the patient's perceived health status.
  A high score corresponds to a better quality of life. The primary endpoint is the difference in total score on the SF-36 at the end of the programme (at 3 months) between the music therapy intervention group and the control group.

SECONDARY OUTCOMES:
Variation of score in the Quality of life assessment (MOS SF-36) | At patient inclusion (V0), at 1 month (V1) and at 3 months from the intervention (V2).
  The variations in the SF-36 quality of life self-assessment scores will be evaluated.
  The repercussions on the quality of life, the anxiety-depressive symptomatology, the well-being at the end of 1 month of intensive music therapy program and at the end of the treatment, at three months will be evaluated.
Hospital Anxiety Depression-Scale (HAD-S) | The evaluations will take place at three times : at baseline (patient inclusion (V0)), at 1 month (V1) and at 3 months from the intervention (V2).
  The HADs is a self-administered questionnaire to identify anxiety and depressive disorders in patients but also in the general population (and not only in hospital practice for which it was originally designed). It is easy to complete and quick to use (completion time: between 2 and 6 minutes).
  For each item, the patient chooses from among the four proposals made, the one that best corresponds to his or her state of mind during the previous week. It consists of 14 items rated from 0 (no symptoms) to 3 according to the severity of the symptoms. Seven questions relate to anxiety and seven to depression, resulting in two scores: A for anxiety and D for depression. The maximum score for each is 21.
  Variations in self-administered scores on perceived anxiety and depressive symptoms of the Hospital Anxiety Depression-Scale (HAD-S) will be evaluated.
Weel-being Scale (EV.I.BE: Echelle d'évaluation instantanée du Bien-Etre) | The evaluations will take place at three times : at baseline (patient inclusion (V0)), at 1 month (V1) and at 3 months from the intervention (V2).
  The EV.I.BE was initially created to assess the perception of quality of life in patients with mild to severe major neurocognitive disorders at a given time. It is a visual analogue scale, i.e. a scale graduated from 1 to 5.
  Variations in the scores obtained on the assessment of well-being using the EV.I.BE (Instantaneous Well-Being Scale) visual analogue scale will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe COUBES, Principal Investigator — Montpellier University Hospital
Locations (1):
- Unité Pathologies Cérébrales Résistantes (UPCR) - Département de Neurochirurgie - Gui de Chauliac, Montpellier, France

REFERENCES:
- [Background] Sihvonen AJ, Sarkamo T, Leo V, Tervaniemi M, Altenmuller E, Soinila S. Music-based interventions in neurological rehabilitation. Lancet Neurol. 2017 Aug;16(8):648-660. doi: 10.1016/S1474-4422(17)30168-0. Epub 2017 Jun 26. PMID 28663005
- [Background] Coubes P, Roubertie A, Vayssiere N, Hemm S, Echenne B. Treatment of DYT1-generalised dystonia by stimulation of the internal globus pallidus. Lancet. 2000 Jun 24;355(9222):2220-1. doi: 10.1016/S0140-6736(00)02410-7. PMID 10881900
- [Background] Ribeiro MKA, Alcantara-Silva TRM, Oliveira JCM, Paula TC, Dutra JBR, Pedrino GR, Simoes K, Sousa RB, Rebelo ACS. Music therapy intervention in cardiac autonomic modulation, anxiety, and depression in mothers of preterms: randomized controlled trial. BMC Psychol. 2018 Dec 13;6(1):57. doi: 10.1186/s40359-018-0271-y. PMID 30545420
- [Background] Hole J, Hirsch M, Ball E, Meads C. Music as an aid for postoperative recovery in adults: a systematic review and meta-analysis. Lancet. 2015 Oct 24;386(10004):1659-71. doi: 10.1016/S0140-6736(15)60169-6. Epub 2015 Aug 12. PMID 26277246
- [Background] Lord VM, Hume VJ, Kelly JL, Cave P, Silver J, Waldman M, White C, Smith C, Tanner R, Sanchez M, Man WD, Polkey MI, Hopkinson NS. Singing classes for chronic obstructive pulmonary disease: a randomized controlled trial. BMC Pulm Med. 2012 Nov 13;12:69. doi: 10.1186/1471-2466-12-69. PMID 23145504